CLINICAL TRIAL: NCT03958708
Title: Modulation of Gut Microbiota by Rifaximin in PD Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chien Tai Hong, Doctor, Assisstant Professor, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201805044
Record Dates: First submitted 2019-05-14; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease; Inflammation
Keywords: gut microbiota; rifaximin
MeSH Terms: conditions — Parkinson Disease; Inflammation | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: People at early stage of Parkinson's disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Rifaximin 550 MG

INTERVENTIONS:
Drug: Rifaximin 550 MG — Rifaximin 550 MG, TWICE A DAY, FOR 7 DAYS

SUMMARY:
The purposes of this clinical trial are to test 1. Whether 1-week rifaximin treatment is able to restore the gut microbiota in a long-term manner in people with Parkinson's disease? 2. Whether the restoration of gut microbiota in people with Parkinson's disease is associated with the reduction of systemic inflammation and circulating exosomal α-synuclein?

DETAILED DESCRIPTION:
Gut microbiota is the largest microorganisms pool in the human body. The physiological roles of gut microbiota for digestion, metabolism, immune homeostasis, GI-tract infection prevention and anti-inflammation. The very first colonized gut microbiota of infant are from maternal vaginal fluid. Gut microbiota are strongly affected by the environment, diet and health status of host.

The alteration of gut microbiota (any microbial imbalance resulting in a shift (i.e., loss or overgrowth of a species) and/or reduction in microbial diversity), which is known as dysbiotic microbiota, is associated with numerous human diseases, including metabolic syndrome, diabetes, obesity, depression and autism. Among people with hypercholesterolemia, they tend to have lower richness and diversity of bacterial communities. In addition, patients with type 2 diabetes were characterized by a moderate degree of gut microbial dysbiosis, a decrease in the abundance of some universal butyrate-producing bacteria and an increase in various opportunistic pathogens, as well as an enrichment of other microbial functions conferring sulphate reduction and oxidative stress resistance. Gut microbiota are also the primary source of short-chain fatty acids (SCFAs). These molecules are known to significantly impact the gut environment and host metabolism and to exhibit potent anti-oxidant and anti-inflammatory properties.

Microbial dysbiosis also impacts on local and systemic inflammation, which are relevant to several human diseases. The gut is the main site for the generation of the two most important T cell populations, the inducible regulatory T cells (iTregs) and CD4IL17-producing cells (Th17). In physiological status, those T cells are responsible for immune tolerance, which avoid inducing immune reaction toward the antigens presented in the gut microbiota9. However, once the detrimental species of gut microbiota trigger the slow and persisted inflammatory process in the gut, intestinal lymphocytes release pro-inflammatory cytokine (IL-1β, IL-6 and TNF), which leads to the elevated intestinal permeability of mucosa. Inflammation induces the permeabilization of gut mucosa and subsequent intestinal leak (leaky gut syndrome). The leaking results in the entrance of large amount of bacterial toxins (such as LPS) into systemic circulation and elevated systemic inflammation.

Gut microbiota also play an important role in several neurological diseases due to the presence of gut-brain axis. Distinct gut microbiota are found in plenty of people with neurological diseases, such as autism, depression, Alzheimer's disease (AD) and Parkinson's disease (PD). Regarding to PD, a neurodegenerative disease with the most well-studied gut-brain axis, 70% people with PD (PwP) suffered from gastrointestinal symptoms and constipation is the most complained. Those symptoms stem from the degeneration of vagus nerve-innervated mesenteric plexus. According to the well-known Braak stage which showed the caudal rostral spreading of Lewy body, medullary vagal nucleus is the first area with the involvement of PD-pathology. In fact, abnormal mesenteric α-synuclein accumulation herald the vagal pathological change. The hypothesis that α-synuclein is originated from intestine is supported by an animal study. Mice with mutated α-synuclein over-expressing had abundant PD-pathology in the midbrain. However, elimination of gut microbiota attenuated the pathology. This study hint that gut microbiota is essential for the aggregation of α-synuclein and the therapeutic potential of modulation gut microbiota for the neuroprotection of PD.

Distinct gut microbiota in PwPs compared with healthy people were demonstrated by several studies: higher level of Akkermansia muciniphila, Bifidobacterium, Methanobrevibacter smithii and Enterobacteriaceae whereas lower level of Prevotellacea, Faecalibacterium prausnitzii and Lactobacilli/Enterococci. Although the causal relationship between PD with the alteration of specific species of bacteria is unknown, some of the bacterial species play role in the aforementioned PD pathogenesis. For instance, Prevotella helps in breaking down complex carbohydrates to produce anti-oxidative, anti-inflammatory SCFAs and neuro-beneficial thiamine and folate and reduce the amount of Prevotella may be harmful for the dopaminergic neurons and augmentation the disease progression.

Modulation of gut microbiota could be achieved by several approaches, such as fecal microbiota transplantation, probiotics and antibiotics. Fecal transplantation obtained certain success in patients with Clostridium difficile infection. In the field of neurological diseases, clinical trials of fecal microbiota transplantation had been launched for children with autism18. However, at the present stage, there is no "standardized" gut microbiota about non-PD people, which limit the application of fecal microbiota transplantation to PwP. Probiotics are easily-available over-the counter supplement which is rich in beneficial micro-organisms. The advantages of probiotics include well-tolerated and minimal adverse effects. Besides, increasing beneficial micro-organisms by intaking probiotics is physiological. However, shared the same disadvantages with fecal microbiota transplantation, there is no specific strain known to be beneficial for PD. Furthermore, comparing with the amount of existing gut microbiota, the probiotics contain far fewer number of micro-organisms. Once the cessation of application, those good micro-organisms are not able to permanently grow in the gut and sometimes even trigger further dysbiosis.

Antibiotics are well-known to modulate the gut microbiota. In fact, the very first time that people are aware of the effect of antibiotics on gut microbiota is the antibiotics-related pseudomembranous colitis, which is secondary to outgrowth of C.difficle due to the loss of normal gut microbiota after the application of potent wide-spectrum antibiotics. Merely all the antibiotics affect gut microbiota more or less, however, the net impact is usually negative. It results in decrease number of beneficial microbiota, increase the harmful strains and reduction the diversity. Unlike the transient effect of probiotics, antibiotics lead to sustained or even permanent alterations. In the clinical observations, the prescription of antibiotics in the childhood is associated with the risk of obesity in the adulthood.

Fortunately, among hundreds of available antibiotics, rifaximin, a non-aminoglycoside semi-synthetic, non-systemic antibiotic derived from rifamycin SV, is known to its unique "eubiotic" effect. Rifaximin is approved by US-FDA in the treatment of traveler's diarrhea and hepatic encephalopathy. According to the literatures, rifaximin did not result in the decrease number of beneficial gut microbiota, such as Lactobacillus and Bifidobacterium. On the other hand, rifaximin did not reduce the diversity of gut microbiota. Most importantly, the effect is long-lasting. The direct effects of rifaximin on pathogens is through reducing the expression of bacterial virulence factors. At the same time, some indirect effects, such as rendering intestinal cells resistant to bacterial colonization, attachment and internalization, and reducing mucosal inflammation work on host.

Instead of the treatment of traveler's diarrhea and hepatic encephalopathy, rifaximin has been applied to PD in clinical trials. PwPs tend to suffer from small intestine bacteria overgrow (SIBO), which affects the absorption of polypeptide, especially levodopa and contributes to the levodopa-induced motor fluctuation. In this trial, prescription of rifaximin, 550mg twice a day for 7 days, significantly reduced the number of undesirable bacteria in the gut, especially H.pylori and improved the response of levodopa. Importantly, the adverse effects are minimal and tolerable1.

At present, there is no available approaches to persistently modulate the gut microbiota of PwPs. Moreover, it is unknown that whether modulate the gut microbiota is beneficial in the clinical and serological biomarkers of PwPs. The present project aims to address these two questions: 1. Whether 1-week rifaximin treatment is able to restore the gut microbiota in a long-term manner in PwPs? 2. Whether the restoration of gut microbiota in PwPs is associated with reduction of systemic inflammation and circulating exosomal α-synuclein?

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease.
2. Hoen and Yahe stage I or II
3. Age between 45-70 years old

Exclusion Criteria:

1. Severe systemic disease (liver cirrhosis greater than Child's A, glomerular filtration rate<60 ml/min/1.73m2, NYHA class 2 and above, or any active malignancy)
2. Past history of following gastrointestinal diseases (inflammatory bowel disease, peptic ulcer with perforation, biliary tract diseases with cholecystectomy, pancreatitis, any gastrointestinal malignancy)
3. Regularly prescribed probiotics or fermented food in past six months
4. Regularly prescribed antibiotics or metformin in the past six months
5. Mini-mental status test below 22 scores.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-05-12 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of gut microbiota | Immediate after treatment/ 6-month after treatment
  Comparing the gut microbiota analyzed by 16sRNA with baseline

SECONDARY OUTCOMES:
Blood biomarkers of neuroinflammation and exosomal alpha-synuclein | 6-month after treatment
  Comparing the blood level of inflammatory/infection markers (TNF-alpha, IL-6, LPS & zonulin) and exosomal alpha-synuclein

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided